CLINICAL TRIAL: NCT03100565
Title: Comparison of Lidocaine Spray With Forced Coughing in Pain Relief During Colposcopy Guided Cervical Biopsy Procedure: A Randomized Controlled Trial
Brief Title: Lidocaine Spray vs Coughing for Pain Relief During Colposcopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, erbil karaman, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YuzuncuYıl
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Colposcopy
Keywords: colposcopy; pain; coughing; anesthetic spray
MeSH Terms: conditions — Pain; Cough

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be blinded to the methods used for pain relief.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colposcopic biopsy under local anesthetic sp (Placebo Comparator)
  Interventions: Drug: local lidocaine spray
- Patients underwent colposcopic biopsy under forced coughing (Placebo Comparator)
  Interventions: Other: forced coughing

INTERVENTIONS:
Drug: local lidocaine spray — The lidocaine spray will be introduced to the cervix just before the biopsy procedure
  Arms: colposcopic biopsy under local anesthetic sp
Other: forced coughing — The patients will be asked to forced coughing during the biopsy procedure
  Arms: Patients underwent colposcopic biopsy under forced coughing

SUMMARY:
Cervical cancer is the third most common genital cancer worldwide. The diagnosis of cervical cancer is performed with the cervical biopsy which is guided by the colposcopy. The colposcopy guided cervical biopsy creates pain and several methods have been reported to overcome the pain related with this procedure. Local anesthetic agent injection into the cervix has been studied and found to be effective and also, forced coughing was compared with local anesthetic injection and it is found to be more effective. In fact local injections can create the pain by itself.However no study compared the effect of forced coughing to local anesthetic spray. The study aims to evaluate the comparison of forced coughing with local anesthetic spray with respect to perceived pain during colposcopy guided biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age >18,
* Presence of cervix,
* Patients who need a diagnostic work up for abnormal cervical smear results.

Exclusion Criteria:

* Pregnancy,
* Presence of already known invasive cancer,
* Allergy to anesthetic agents.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Pain during procedure evaluated by the 0-10 cm scale of Visual analog scale (VAS) scoring system | 0-1 min
  The perceived pain will be measured during the biopsy procedure. It will be evaluated by the 0-10 cm scale of VAS scoring system. The patient will be asked to rate her pain as 0 corresponds ''no pain'' and 10 to the '' worst pain''

SECONDARY OUTCOMES:
Pain at the 30th minutes after the procedure evaluated by the 0-10 cm scale of VAS scoring system | 30. Min
  The perceived pain will be measured after the biopsy procedure (at the 30th min). It will be evaluated by the 0-10 cm scale of VAS scoring system. The patient will be asked to rate her pain as 0 corresponds ''no pain'' and 10 to the '' worst pain''

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Medical faculty, department of obstetric and gynecology, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No